CLINICAL TRIAL: NCT04755816
Title: A Multifaceted Adaptive Mobile Application to Promote Self-management and Improve Outcomes in Heart Failure
Brief Title: A Mobile Application to Promote Self-management and Improve Outcomes in Heart Failure
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow recruitment - DSMB decision
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Michael Dorsch, Associate Professor of Clinical Pharmacy, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HUM00181316; R01AG062582-01A1 (NIH)
Record Dates: First submitted 2021-01-27; First posted 2021-02-16 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group 'A' (Sham Comparator): Standard heart failure educational information.
  Interventions: Behavioral: Educational content
- Dietary Sodium Intervention 'B' (Experimental): The dietary sodium intervention facilitates lower sodium choices using tailored push notifications.
  Interventions: Behavioral: Sodium intervention
- Clinical Worsening Intervention 'C' (Experimental): The clinical worsening intervention promotes self-monitoring and self-management and is linked tailored push notifications.
  Interventions: Behavioral: Clinical worsening intervention
- Dietary Sodium and Clinical Worsening 'D' (Experimental): Full access to all content in the control, dietary sodium, and clinical worsening interventions.
  Interventions: Behavioral: Sodium intervention; Behavioral: Clinical worsening intervention

INTERVENTIONS:
Behavioral: Sodium intervention — The sodium dietary intervention provides the user with a tailored message to assist with making dietary choices based on sodium content when they arrive at a grocery store or restaurant.
  Arms: Dietary Sodium Intervention 'B'; Dietary Sodium and Clinical Worsening 'D'
Behavioral: Clinical worsening intervention — The intervention adapts to the participant's reported symptoms and provides feedback with a global health status indicator (HSI). Users will receive tailored push notification based on their HSI status.
  Arms: Clinical Worsening Intervention 'C'; Dietary Sodium and Clinical Worsening 'D'
Behavioral: Educational content — Standard heart failure educational information and a daily symptom survey.
  Arms: Control Group 'A'

SUMMARY:
This study will investigate the effectiveness of two contextual just-in-time adaptive interventions (JITAIs) delivered via a mobile app for heart failure patients.

DETAILED DESCRIPTION:
The Manage HF study is a multicenter 12-week randomized controlled double-blind 2x2 factorial clinical trial. This study will investigate the effectiveness of two contextual just-in-time adaptive interventions (JITAIs) delivered via a mobile app for heart failure patients. The clinical worsening intervention targets self-management of behaviors to prevent worsening of a patient's heart failure symptoms. The dietary sodium intervention promotes lower sodium intake. Eligible participants will be randomized to the dietary sodium intervention, the clinical worsening intervention, both interventions, or no intervention in a 1:1:1:1 manner, stratified by site, gender, and HF type (HFpEF versus HFrEF).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older at screening
2. Currently admitted or discharged from the hospital within the last 14 days with a diagnosis of acute or acute on chronic decompensated HF.
3. Based on one of the EF criteria (LVEF within 12 months of randomization. BNP or NT-proBNP criteria within 30 days prior to randomization):

   * Left ventricular ejection fraction (LVEF) ≤ 40%.
   * LVEF >40% and BNP > 175 pg/ml or NT-proBNP > 700 pg/ml. Thresholds for NT-proBNP and BNP for LVEF > 40% will be corrected for body mass index (BMI) using a 4% reduction per BMI unit over 25 kg/m2.
4. Have a personal physician for follow-up
5. A smartphone with a compatible Apple or Android operating system installed and able to download and use ManageHF including accepting all permissions
6. A valid email address
7. Fluent in spoken and written English

Exclusion Criteria:

1. Contraindication to recommending a sodium restriction diet
2. Scheduled intervention for primary valvular heart disease will occur during the study period.
3. Cardiac resynchronization therapy (CRT) within 3 months prior to screening or current plan to implant CRT device during the study period.
4. Dialysis
5. Previous cardiac transplantation or implantation of a ventricular assistance device or similar device.
6. Listed status 1, 2 or 3 for heart transplant
7. Implantation of a ventricular assistance device is expected within 3 months after randomization
8. Non-cardiac illness with expected survival of less than 3 months
9. Discharge to a setting other than home
10. Requirement for chronic inotropic therapy (e.g. milrinone, dobutamine)
11. Inability to use Withings devices due to equipment limitations or contraindications
12. Currently pregnant or intend to become pregnant during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dorsch, PharmD, Principal Investigator — University of Michigan
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Stanford, California
  - Emory University, Atlanta, Georgia
  - Atlanta VA Health Care System, Decatur, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital System, Detroit, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
The aim is to prepare data for deposit into the National Institute on Aging supported National Archive of Computerized Data on Aging data repository. The de-identified analytic data will be prepared as SAS transport files or ASCII comma-delimited files with accompanying codebooks that describe the data and data structure. The redaction will employ best practices and will be consistent with National Institute on Aging data sharing policies.
Supporting Information: Study Protocol, ICF
Time Frame: No later than 3 years after the end of the study or 2 years after the main paper reporting the results of the trial, whichever comes first.
Access Criteria: Researchers at institutions with a Federal Wide Assurance will be able to gain access to repository data by submitting a data access request in accordance with applicable policies.

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Standard heart failure educational information.
  Educational content: Standard heart failure educational information and a daily symptom survey.
- Dietary Sodium Intervention: The dietary sodium intervention facilitates lower sodium choices using tailored push notifications.
  Sodium intervention: The sodium dietary intervention provides uses location services to determine when a participant is at home, arrives at a grocery store or arrives at a restaurant. The user receives a tailored message to assist with making dietary choices based on sodium content.
- Clinical Worsening Intervention: The clinical worsening intervention promotes self-monitoring and self-management and is linked tailored push notifications.
  Clinical worsening intervention: The intervention adapts to the participant's reported symptoms and provides feedback with a global health status indicator (HSI). Users will receive tailored push notification based on their HSI status.
- Dietary Sodium and Clinical Worsening: Full access to all content in the control, dietary sodium, and clinical worsening interventions.
  Sodium intervention: The sodium dietary intervention provides uses location services to determine when a participant is at home, arrives at a grocery store or arrives at a restaurant. The user receives a tailored message to assist with making dietary choices based on sodium content.
  Clinical worsening intervention: The intervention adapts to the participant's reported symptoms and provides feedback with a global health status indicator (HSI). Users will receive tailored push notification based on their HSI status.
Period: Overall Study
Arm/Group | Control Group | Dietary Sodium Intervention | Clinical Worsening Intervention | Dietary Sodium and Clinical Worsening
Started | 12 | 20 | 12 | 18
Completed | 12 | 20 | 12 | 18
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Dietary Sodium Intervention | Clinical Worsening Intervention | Dietary Sodium and Clinical Worsening | Total
Number analyzed (Participants) | 12 | 20 | 12 | 18 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 16 | 10 | 12 | 46
  >=65 years | 4 | 4 | 2 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (13.04) | 54.1 (15.6) | 54 (11.53) | 54.8 (16.6) | 54.8 (14.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 4 | 6 | 20
  Male | 9 | 13 | 8 | 12 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 11 | 19 | 12 | 18 | 60
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 7 | 13 | 7 | 7 | 34
  White | 4 | 6 | 5 | 10 | 25
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Hierarchical Combination ("Win Ratio") of Time to All-cause Mortality, Time to Heart Failure Hospital Readmission, and Decline in Health-related Quality of Life (HRQOL) [ Time Frame: Baseline up to Week 12 ]
Description: Time to all-cause mortality (ACM), time to heart failure hospital readmission (HFHR), and decline in quality of life will be analyzed using the Finkelstein-Schoenfeld method. The method combines these three endpoints in a hierarchical fashion using ACM first, HRHR second, and change in HRQOL third. The method pairs every participant receiving the diet intervention with every participant not receiving the diet intervention within each stratum. Within each pairing, a +1 is assigned to the "better" participant, -1 to the "worse" participant, and 0 if they are "tied". The comparison begins with ACM. Tied pairings are then compared using HFHR. Any remaining tied pairings are compared using change in HRQOL. A 'Win' represents a participant doing better within each pairing (receiving +1) based on the hierarchical comparison. The reported unit is the total "wins" for each intervention group from performing such a hierarchical comparison across all strata.
Time Frame: 12 weeks
Population: Subjects randomized to the Dietary intervention only (n=20) + those randomized to both interventions (n=18) vs Subjects randomized to the Clinical Worsening intervention only (n=12) + those randomized to Neither intervention (n=12)
Measure: Number; unit: Total number of wins
Groups:
- Dietary Sodium Intervention: The sodium dietary intervention provides the user with tailored messages to assist with making dietary choices based on sodium content when they arrive at a grocery store or a restaurant.
  This includes group B and D.
- No Dietary Sodium Intervention: Access to all content in the control, and clinical worsening interventions. This includes group A and C.
Arm/Group | Dietary Sodium Intervention | No Dietary Sodium Intervention
Number analyzed (Participants) | 38 | 24
Total number of wins
  Time to All-Cause Death | 0 | 0
  Time to Heart-Failure Readmission | 136 | 156
  Change in MLHFQ from Baseline to 12 Weeks | 146 | 63
  Overall (across 3 outcomes) | 282 | 219
Statistical Analysis 1: Comparison: Dietary Sodium Intervention vs No Dietary Sodium Intervention; Dietary Sodium Intervention includes those in treatment group B and D. No Dietary Sodium Intervention includes those in treatment group A and C. By the unmatched pairs win ratio method, each participant receiving the intervention will be compared to each participant not receiving the intervention. For each comparison, "winners" will be determined according to the hierarchy described above. The win ratio is the number winners divided by the number of losers associated with the intervention."; Test type: Other — Estimates and confidence intervals are provided; Win Ratio = 1.29, 95% CI 2-sided [1.08 to 1.54]

2. Primary Outcome: Hierarchical Combination ("Win Ratio") of Time to All-cause Mortality, Time to Heart Failure Hospital Readmission, and Decline in Health-related Quality of Life (HRQOL) [ Time Frame: Baseline up to Week 12 ]
Description: Time to all-cause mortality (ACM), time to heart failure hospital readmission (HFHR), and decline in quality of life will be analyzed using the Finkelstein-Schoenfeld method. The method combines these three endpoints in a hierarchical fashion using ACM first, HRHR second, and change in HRQOL third. The method pairs every participant receiving the clinical worsening intervention with every participant not receiving the clinical worsening intervention within each stratum. Within each pairing, a +1 is assigned to the "better" participant, -1 to the "worse" participant, and 0 if they are "tied". The comparison begins with ACM. Tied pairings are then compared using HFHR. Any remaining tied pairings are compared using change in HRQOL. A 'Win' represents a participant doing better within each pairing (receiving +1) based on the hierarchical comparison. The reported unit is the total "wins" for each intervention group from performing such a hierarchical comparison across all strata.
Time Frame: 12 weeks
Population: Subjects randomized to the Clinical Worsening intervention only (n=12) + those randomized to both interventions (n=18) vs Subjects randomized to the Dietary intervention only (n=20) + those randomized to Neither intervention (n=12)
Measure: Number; unit: Total number of wins
Groups:
- Clinical Worsening Intervention: Access to all content in the dietary sodium, and clinical worsening interventions. This includes group C and D.
  Sodium intervention: The sodium dietary intervention provides uses location services to determine when a participant is at home, arrives at a grocery store or arrives at a restaurant. The user receives a tailored message to assist with making dietary choices based on sodium content.
  Clinical worsening intervention: The intervention adapts to the participant's reported symptoms and provides feedback with a global health status indicator (HSI). Users will receive tailored push notification based on their HSI status.
- No Clinical Worsening Intervention: Access to all content in the control, and dietary sodium. This includes group A and B.
  Educational content: Standard heart failure educational information and a daily symptom survey.
  Sodium intervention: The sodium dietary intervention provides uses location services to determine when a participant is at home, arrives at a grocery store or arrives at a restaurant. The user receives a tailored message to assist with making dietary choices based on sodium content.
Arm/Group | Clinical Worsening Intervention | No Clinical Worsening Intervention
Number analyzed (Participants) | 30 | 32
Total number of wins
  Time to All-Cause Death | 0 | 0
  Time to Heart-Failure Readmission | 136 | 156
  Change in MLHFQ from Baseline to 12 Weeks | 146 | 63
  Overall (across 3 outcomes) | 282 | 219
Statistical Analysis 1: Comparison: Clinical Worsening Intervention vs No Clinical Worsening Intervention; Clinical Worsening Intervention includes those in treatment group C and D. No Clinical Worsening Intervention includes those in group A and B. By the unmatched pairs win ratio method, each participant receiving the intervention will be compared to each participant not receiving the intervention. For each comparison, "winners" will be determined according to the hierarchy described above. The win ratio is the number winners divided by the number of losers associated with the intervention."; Test type: Other — Estimates and confidence intervals are provided; Win Ratio = 1.29, 95% CI 2-sided [1.08 to 1.54]

3. Secondary Outcome: All-Cause Mortality [ Time Frame: Baseline up to Week 12 ]
Description: Time to all-cause mortality will be analyzed up to week 12.
Time Frame: 12 weeks
Population: no deaths in the study and this outcome could not be assessed
Arm/Group | Control Group | Dietary Sodium Intervention | Clinical Worsening Intervention | Dietary Sodium and Clinical Worsening
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Heart Failure-related Hospitalizations [ Time Frame: Baseline up to Week 12 ]
Description: Time to first heart-failure related hospitalization will be analyzed up to week 12.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days since randomization
Groups:
- No Dietary Sodium Intervention: Access to all content in the control, and clinical worsening interventions. Includes group A and C.
Arm/Group | Dietary Sodium Intervention | No Dietary Sodium Intervention
Number analyzed (Participants) | 38 | 24
Days since randomization | 43.4285714 (24.4871200) | 48.5000000 (19.3649167)
Statistical Analysis 1: Comparison: Dietary Sodium Intervention vs No Dietary Sodium Intervention; Dietary Sodium Intervention includes those in treatment group B and D. No Dietary Sodium Intervention includes those in treatment group A and C; Test type: Other — Estimates and confidence intervals are provided; Hazard Ratio (HR) = 1.096, 95% CI 2-sided [0.321 to 3.743]

5. Secondary Outcome: Change From Baseline in Health-related Quality of Life [ Time Frame: Baseline up to Week 12 ]
Description: Change from baseline to week 12 in health-related quality of life as measured by the Minnesota Living with Heart Failure Questionnaire.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on MLHFQ scale
Arm/Group | Dietary Sodium Intervention | No Dietary Sodium Intervention
Number analyzed (Participants) | 27 | 12
Points on MLHFQ scale | -39.70 (33.908) | -24.33 (24.828)
Statistical Analysis 1: Comparison: Dietary Sodium Intervention vs No Dietary Sodium Intervention; Dietary Sodium Intervention includes those in treatment group B and D. No Dietary Sodium Intervention includes those in treatment group A and C. Simple linear regression models will be used to assess the outcome of change in MLHFQ over 12 weeks as a function of treatment group assignment. Beta coefficients and 95% confidence intervals will be reported; Test type: Other — Estimates and confidence intervals are provided; Slope = -15.37, 95% CI 2-sided [-37.5 to 6.76] — The total score for the MLHFQ ranges from 0 to 105, with higher scores indicating more significant impairment in health-related quality of life. "The change in MLHFQ is defined as MLHFQ at Week 12 minus MLHFQ at Week 0."

6. Secondary Outcome: Heart Failure-related Hospitalizations [ Time Frame: Baseline up to Week 12 ]
Description: Time to first heart-failure related hospitalization will be analyzed up to week 12.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days since randomization
Arm/Group | Clinical Worsening Intervention | No Clinical Worsening Intervention
Number analyzed (Participants) | 30 | 32
Days since randomization | 53.7500000 (14.4308697) | 40.4285714 (24.8720535)
Statistical Analysis 1: Comparison: Clinical Worsening Intervention vs No Clinical Worsening Intervention; Clinical Worsening Intervention includes those in treatment group C and D. No Clinical Worsening Intervention includes those in treatment group A and B; Test type: Other — Estimates and confidence intervals are provided; Hazard Ratio (HR) = 0.556, 95% CI 2-sided [0.163 to 1.901]

7. Secondary Outcome: Change From Baseline in Health-related Quality of Life [ Time Frame: Baseline up to Week 12 ]
Description: as for outcome 5
Time Frame: 12 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Points on MLHFQ scale
Arm/Group | Clinical Worsening Intervention | No Clinical Worsening Intervention
Number analyzed (Participants) | 17 | 22
Points on MLHFQ scale | -42.29 (28.169) | -29.32 (34.036)
Statistical Analysis 1: Comparison: Clinical Worsening Intervention vs No Clinical Worsening Intervention; Clinical Worsening Intervention includes those in treatment group C and D. No Clinical Worsening Intervention includes those in treatment group A and B. Simple linear regression models will be used to assess the outcome of change in MLHFQ over 12 weeks as a function of treatment group assignment. Beta coefficients and 95% confidence intervals will be reported; Test type: Other — Estimates and confidence intervals are provided; Slope = -12.98, 95% CI 2-sided [-33.67 to 7.72] — [estimate comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: The adverse event data were collected from September of 2021 to June of 2022, so a total of 9 months. Each participants was assessed for AEs for the follow-up period of 12 weeks from baseline.
Description: The number of participants at risk for All-Cause Mortality is zero because there were no deaths reported in the study.
Arm/Group | Control Group | Dietary Sodium Intervention | Clinical Worsening Intervention | Dietary Sodium and Clinical Worsening
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/20 | 0/12 | 0/18
Serious Adverse Events (participants affected / at risk) | 5/12 | 9/20 | 4/12 | 6/18
Other Adverse Events (participants affected / at risk) | 3/12 | 4/20 | 3/12 | 2/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group (N=12) | Dietary Sodium Intervention (N=20) | Clinical Worsening Intervention (N=12) | Dietary Sodium and Clinical Worsening (N=18)
Inpatient hospitalization or prolongation of existing hospitalization (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 — SAE were not monitored with regard to specific adverse event terms
Inpatient hospitalization or prolongation of existing hospitalization (Cardiac disorders) | 2 | 5 | 2 | 1 — SAE were not monitored with regard to specific adverse event terms
Inpatient hospitalization or prolongation of existing hospitalization (Endocrine disorders) | 1 | 1 | 0 | 0 — SAE were not monitored with regard to specific adverse event terms
Inpatient hospitalization or prolongation of existing hospitalization (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — SAE were not monitored with regard to specific adverse event terms
Inpatient hospitalization or prolongation of existing hospitalization (Infections and infestations) | 0 | 1 | 0 | 0 — SAE were not monitored with regard to specific adverse event terms
Inpatient hospitalization or prolongation of existing hospitalization (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 — SAE were not monitored with regard to specific adverse event terms
Inpatient hospitalization or prolongation of existing hospitalization (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 — SAE were not monitored with regard to specific adverse event terms
Inpatient hospitalization or prolongation of existing hospitalization (Investigations) | 0 | 0 | 0 | 1 — As other. SAE were not monitored with regard to specific adverse event terms
Inpatient hospitalization or prolongation of existing hospitalization (Psychiatric disorders) | 0 | 1 | 0 | 0 — SAE were not monitored with regard to specific adverse event terms
Inpatient hospitalization or prolongation of existing hospitalization (Renal and urinary disorders) | 1 | 0 | 0 | 2 — SAE were not monitored with regard to specific adverse event terms
Inpatient hospitalization or prolongation of existing hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 — SAE were not monitored with regard to specific adverse event terms
Life Threatening (Cardiac disorders) | 0 | 0 | 0 | 1 — SAE were not monitored with regard to specific adverse event terms
Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 — SAE were not monitored with regard to specific adverse event terms
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group (N=12) | Dietary Sodium Intervention (N=20) | Clinical Worsening Intervention (N=12) | Dietary Sodium and Clinical Worsening (N=18)
Hyperkalemia (Potassium > 6.0 meq/dl or requiring change in therapy) (Renal and urinary disorders) | 1 | 0 | 0 | 0
Symptomatic bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Symptomatic hypotension (Blood and lymphatic system disorders) | 1 | 1 | 2 | 0
Worsening renal function (increase in creatinine by 0.5 mg/dl from last visit or requiring change in (Renal and urinary disorders) | 0 | 3 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/16/NCT04755816/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/16/NCT04755816/SAP_001.pdf
  • Informed Consent Form (2022-04-23): https://cdn.clinicaltrials.gov/large-docs/16/NCT04755816/ICF_002.pdf